CLINICAL TRIAL: NCT03271372
Title: A Multicenter, Randomized, Double-Blinded, Placebo-Controlled, Phase 3 Trial of Adjuvant Avelumab (Anti-PDL-1 Antibody) in Merkel Cell Carcinoma Patients With Lymph Node Metastases
Brief Title: Adjuvant Avelumab in Merkel Cell Cancer
Acronym: ADAM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9820; NCI-2017-00998 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1717054 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Stage III Merkel Cell Carcinoma AJCC v8; Stage IIIB Merkel Cell Carcinoma AJCC v8; Stage IIIA Merkel Cell Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — avelumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (avelumab) (Experimental): Patients receive avelumab IV over 1 hour once every 15 days for the first 120 days (Induction Phase 1), once every 30 days for the next 120 days (Induction Phase 2), and then once every 120 days (Maintenance Phase) for a maximum of 720 days (approximately 24 months or 2 years total) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Other: Peripheral Blood Collection
- Arm II (placebo) (Placebo Comparator): Patients receive placebo IV over 1 hour once every 15 days for the first 120 days (Induction Phase 1), once every 30 days for the next 120 days (Induction Phase 2), and then once every 120 days (Maintenance Phase) for a maximum of 720 days (approximately 24 months or 2 years total) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Peripheral Blood Collection; Other: Placebo

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
  Arms: Arm I (avelumab)
Other: Peripheral Blood Collection — Correlative studies
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; normal saline solution
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase III trial studies how well avelumab works in treating patients with Merkel cell cancer that has spread to the lymph nodes and have undergone surgery and/or radiation therapy. Immunotherapy with monoclonal antibodies, such as avelumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
OUTLINE:

Patients are randomized to 1 of 2 arms.

ARM I: Patients receive avelumab intravenously (IV) over 1 hour once every 15 days for the first 120 days (Induction Phase 1), once every 30 days for the next 120 days (Induction Phase 2), and then once every 120 days (Maintenance Phase) for a maximum of 720 days (approximately 24 months or 2 years total) in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo IV over 1 hour once every 15 days for the first 120 days (Induction Phase 1), once every 30 days for the next 120 days (Induction Phase 2), and then once every 120 days (Maintenance Phase) for a maximum of 720 days (approximately 24 months or 2 years total) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 5 years from day 1 and then once every 12 months until the study is terminated by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed MCC metastases in regional lymph node(s)

  * Confirmation of the MCC diagnosis in the regional lymph node(s) is mandatory for trial participation
  * (NOTE: In-transit metastases without regional nodal involvement could be allowed, but only after written approval of the medical monitor)
* Must have completed definitive treatment for primary MCC and regional lymphatic metastases that included surgical removal (with/without adjuvant radiation therapy) or primary radiation therapy as determined by the treating investigator
* Aged >= 18 years. Both men and women, and members of all races and ethnic groups are eligible for this trial.
* Estimated life expectancy greater than 3 years
* Must start the study treatment no more than 120 days from the start date of definitive therapy (the date of surgical removal of nodal metastases or the date of initiation of definitive radiation therapy, as applicable)
* Eastern Co-Operative Group (Eastern Cooperative Oncology Group [ECOG]) performance score of 0 or 1
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 9 g/dL (may have been transfused)
* Total bilirubin level ≤ 1.5 x the upper limit of normal (ULN) range
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 x ULN
* Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula or by 24-hour urine collection for creatinine clearance or according to local institutional standard
* Women of childbearing potential must have a negative serum or urine pregnancy test at screening
* Both male and female subjects must be willing to use highly effective contraception (that is, methods with a failure rate of less than 1% per year) throughout the study and for at least 30 days after last avelumab treatment administration if the risk of conception exists

  * (NOTE: The effects of the study treatment on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use highly effective contraception, as stipulated in national or local guidelines. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the treating physician should be informed immediately.)
* Must have an ability to understand and the willingness to sign a written informed consent document
* Must consent to allow the acquisition of existing formalin-fixed paraffin-embedded (FFPE) tumor tissue, either a block or unstained slides, for performance of correlative studies

Exclusion Criteria:

* Clinical or radiologic suspicion of residual MCC at the time of enrollment
* Suspicion or known history of distant metastatic MCC, which is not classifiable as local recurrence or regional metastasis
* Any prior systemic therapy (e.g. adjuvant, neo-adjuvant or concurrent use of chemotherapy, immunotherapy or an investigational agent) for MCC at any time
* Any prior intra-lesional MCC therapy within 180 days from day 1 of study treatment
* Residual toxicity from prior therapy grade > 1 (National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [NCI-CTCAE v 5.0]) that could interfere with study endpoints or put patient safety at risk
* Previous malignant disease (other than Merkel cell carcinoma) diagnosed within 3 years from day 1 of study treatment that could interfere with study endpoints or put patient safety at risk

  * (NOTE: Exception will be made for adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ [skin, bladder, cervical, colorectal, breast] or low grade prostatic intraepithelial neoplasia or Grade 1 prostate cancer; any other neoplasm, which is adjudged by the treating investigator to have a low risk of recurrence during the study, could be enrolled only after written approval from the medical monitor)
* Use of any systemic immunosuppressive treatments including corticosteroids, cyclosporine, mycophenolate mofetil et cetera, ongoing or within the last 3 months prior to day 1 of treatment

  * (NOTE: Patients on physiologic dose of corticosteroids [≤ 10 mg/day of prednisone or equivalent] for long-term hormone-replacement therapy or those requiring short, intermittent courses of corticosteroids for hypersensitivity prophylaxis [such as for iodinated computed tomography (CT) contrast prophylaxis] or those using intranasal, inhaled, topical steroids, or local steroid injection [e.g., intra-articular injection] can be allowed)
* Immunosuppressed status due to known human immunodeficiency virus (HIV) infection, severe uncontrolled diabetes, concurrent hematological malignancy, or other comorbidities
* Uncontrolled intercurrent illness including, but not limited to, active serious infection, active hepatitis B or hepatitis C infection, uncontrolled seizure disorder, substance abuse disorder, or psychiatric illness/social situations that would limit compliance with study requirements or would put the patient at increased risk of complications during the study period
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
* Active or history of any serious autoimmune disease, prior organ transplantation, including allogeneic stem-cell transplantation or immune-deficiencies that required treatment with systemic immunosuppressive drugs and could flare-up during study treatment

  * (NOTE: Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible)
* Other severe acute or chronic medical conditions including immune-mediated colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Known prior severe hypersensitivity to investigational product or any component in its formulations that could interfere with study endpoints or put patient safety at risk
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2029-02-18 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | From the date of randomization and the date of first recurrence or death (whatever the cause), whichever occurs first, assessed for up to 5 years
  The Kaplan-Meier technique will be used to obtain estimates.

SECONDARY OUTCOMES:
Overall survival | From the date of randomization and the date of death, assessed for up to 5 years then every 12 months after study drug discontinued
  The Kaplan-Meier technique will be used to obtain estimates.
Disease-specific survival | From the date of randomization and the date of death from Merkel cell carcinoma, assessed for up to 5 years
  Cumulative incidence estimates will be used to summarize the probabilities of disease-specific survival.
Distant-metastases free survival | From the date of randomization and the date of first distant metastasis or date of death (any cause), whichever occurs first, assessed for up to 5 years
  The Kaplan-Meier technique will be used to obtain estimates.
Incidence of adverse events | Throughout the duration of the treatment (up to 2 years after randomization)
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.

OTHER OUTCOMES:
AMERK serology | Up to 5 years
  Blood test to predict recurrence in those patients who had a positive titer at baseline.
Biomarker exploration in tumor and peripheral blood samples | Up to 5 years
  Tumor and peripheral blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Shailender Bhatia, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (9):
- United States (9):
  - University of California Irvine Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No